CLINICAL TRIAL: NCT04952571
Title: An Exploratory Study on Camrelizumab Combined with Bevacizumab for Adult Patients with Recurrent Glioblastoma (GBM)
Brief Title: Combined Treatment of Camrelizumab and Bevacizumab for Adult Patients with Recurrent Glioblastoma (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Beijing Sanbo Brain Hospital, Beijing Sanbo Brain Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-GBM-II-007
Record Dates: First submitted 2021-06-23; First posted 2021-07-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Glioblastoma
Keywords: Recurrent Glioblastoma; Immunotherapy; antiangiogenesis
MeSH Terms: conditions — Glioblastoma | interventions — camrelizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: glioblastoma at first relapse, glioblastoma at second relapse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GBM at first relapse (Experimental)
  Interventions: Drug: Camrelizumab and Bevacizumab
- GBM at second relapse (Experimental)
  Interventions: Drug: Camrelizumab and Bevacizumab

INTERVENTIONS:
Drug: Camrelizumab and Bevacizumab — Stage 1: Targeted therapy induction phase: bevacizumab 5mg/kg, intravenous infusion, once every two weeks, 2 cycles in total.
  Phase 2: Targeted combined immunotherapy: once every three weeks with the following drugs: (1) bevacizumab 7.5mg/kg intravenously;(2) Carrelizumab: 200mg/ time, intravenous infusion.

SUMMARY:
This study is intend to explore the efficacy and safety of combined treatment of camrelizumab and bevacizumab in adult patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
There is no effective chemotherapy regimen for recurrent glioblastoma. The antiangiogenic drug bevacizumab has high objective response rate and rapid onset, but the duration of efficacy needs to be improved.The objective response rate of PD-1 monoclonal antibody immunotherapy is low and the onset of the effect is slow, but the effective patients have a long duration of efficacy.The combined treatment of PD-1 monoclonal antibody and bevacizumab may learn from each other to improve the effective rate, shorten the onset time and prolong the duration of efficacy.Studies have shown that bevacizumab can enhance the efficacy of immunotherapy in a variety of cancers, including melanoma, kidney cancer, non-small cell lung cancer, and liver cancer.However, previous studies have shown limited efficacy of PD-1 monoclonal antibody combined with bevacizumab in the treatment of recurrent glioblastoma.

In this study, the combination therapy was optimized by introducing induction phase therapy, which is expected to further improve the efficacy. In our previous exploratory treatment of patients with severe recurrent glioblastoma after multiple treatments, the initial efficacy was considerable.

The purpose of this study is to evaluate the efficacy and safety of camrelizumab [a programmed cell death 1 (PD-1) inhibitor] combined with bevacizumab for adult patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~70, male or female
2. Primary supratentorial glioblastoma with first or second rogression/recurrence
3. IDH1/2 wildtype
4. KPS score ≥70 in patients with the first recurrence and ≥60 in patients with the second recurrence
5. Expected survival ≥12 weeks.
6. The time interval from the last radiotherapy was ≥12 weeks, unless there was new tumor enhancement in the radiological field or clear evidence of tumor hipathology.
7. Radiotherapy and at least one regimen of chemotherapy before recurrence (excluding temozolomide chemotherapy during concurrent radiotherapy).
8. The patients were enrolled after the end of the previous chemotherapy interval and had recovered from the related adverse reactions (except hair loss and pigmentation).
9. The tumor was confirmed to have definite recurrence by MRI, with enhanced lesion diameter ≥1cm and ≥2 layers (layer spacing 5mm), or was confirmed to have recurrence by pathology after re-biopsy or surgery.
10. The time interval between the last operation and the last biopsy was ≥4 weeks or ≥2 weeks at the time of enrollment.
11. The main organs function normally, no serious abnormal blood, heart, lung, liver, kidney function and immune deficiency diseases
12. Women of childbearing age are required to have a negative pregnancy test (serum or urine) within 7 days before enrolment and to voluntarily use contraception during treatment and within 8 weeks after the last treatment;For men, they should be surgically sterilized or agree to use contraception during treatment and for 8 weeks after the last treatment.
13. Patients voluntarily enrolled in this study and signed informed consent (ICF).
14. Good compliance is expected, efficacy and adverse reactions can be followed up according to protocol requirements

Exclusion Criteria:

1. Glioblastoma in the midline (thalamus, brainstem, sellar region, etc.).
2. Patients with initial recurrence had previously received long-term high-dose antiangiogenic drugs (except those with amlotinib or apatinib for less than 1 month and no progress during treatment, except those with intermittent bev dose intensity ≤5mg/ week and ≤3 times) or immunocheckpoint inhibitors, TCR-T, CAR-T, etc.;Patients with secondary recurrence had previously received long-term high-dose therapy of Bev (except for intermittent Bev dose intensity ≤5mg/ week and ≤3 times) or immunocheckpoint inhibitors, TCR-T, or CAR-T.
3. Other study drugs are being used.
4. An allergic reaction or intolerance to any component of the drug used in this study is known.
5. Other malignant tumors in the past 3 years.
6. Subjects who had been systematically treated with corticosteroids (>4mg/day dexamethasone or other equivalent hormone) or other immunosuppressants within 2 weeks prior to first use of carrelizumab.In the absence of active autoimmune disease, inhaled or topical corticosteroids and hormone replacement therapy with doses less than or equal to 4mg/ day of dexamethasone are permitted.
7. The presence or history of any active autoimmune disease .
8. Uncontrolled hypertension.
9. Myocardial infarction occurred within 6 months prior to enrollment, New York Heart Society Class II heart failure or above, uncontrolled angina pectoris, uncontrolled severe arrhythmias, clinically significant pericardial disease, and electrocardiogram indicating acute ischemia or abnormal active conduction system.
10. Abnormal coagulation function, bleeding tendency or receiving thrombolytic or anticoagulant therapy.
11. Before entering the study 3 months there have been significant clinical significance of bleeding symptoms or have definite bleeding tendency;Or arterial/venous thrombosis events, such as cerebrovascular accidents, deep vein thrombosis and pulmonary embolism, occurred within 6 months before the study.
12. Severe infection occurred within 4 weeks prior to initial administration;Or unexplained fever >38.5℃ during screening/prior to first administration.
13. People who have a history of abuse of psychotropic substances and are unable to get rid of them or have mental disorders.
14. Had major surgery or had an open wound or fracture within 4 weeks prior to first administration.
15. Empty sinus passages or perforations were observed within 6 months prior to study entry.
16. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBVDNA≥500IU/ mL), hepatitis C (positive hepatitis C antibody and HCV-RNA above the detection limit of the assay method) or co-infection with hepatitis B and hepatitis C.
17. Patients who received anti-tumor vaccine or other immunomodulatory drugs within 4 weeks before enrolment;Patients who have received or will receive live attenuated or recombinant vaccine within 4 weeks;Patients who received or will receive the inactivated vaccine within 1 week.
18. Pregnancy and lactation.
19. Other conditions that the investigator considered inappropriate for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | Up to three years
  Progression-free survival rate at 6 months

SECONDARY OUTCOMES:
OS(overall survival) | Up to three years
  the time interval from entry to death from any cause or last follow-up and is measured in the intent-to-treat population
PFS(progression free survival) | Up to three years
  the time interval from entry to tumor progression, death from any cause, or last follow-up
ORR(objective response rate) | Up to three years
  rate of CR+PR
DCR（Disease Control Rate） | Up to three years
  rate of CR+PR+SD
The correlation between KPS change and efficacy | Up to three years
  the correlation between KPS baseline, KPS change (increase, decrease,stable) and best efficacy (CR, PR, SD, PD).
Median duration of KPS ≥ 70 | Up to three years
  Median duration of KPS ≥ 70 during progression-free survival
Frequency and severity of treatment-related adverse events | Up to three years
  Frequency and severity of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Median duration of stable/improved quality of life assessed by EORTC QLQ-C30 | Up to three years
  the time interval from entry to change of ≥10 points on the EORTC QLQ-C30 without further improvement or disease progression or death.
Median duration of stable/improved quality of life assessed by EORTC QLQ-BN20 | Up to three years
  the time interval from entry to change of ≥10 points on the EORTC QLQ-BN20 without further improvement or disease progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sanbo Brain Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No